CLINICAL TRIAL: NCT04376086
Title: Segmental Epidural Block for Feeding Jejunostomy in Cancer Patients
Brief Title: Segmental Epidural Block for Feeding Jeujunostomy in Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Walaa Youssef Elsabeeny, Lecturer of anesthesia and pain management, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AP1904-50103
Record Dates: First submitted 2020-04-10; First posted 2020-05-06 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Anesthesia
MeSH Terms: interventions — Anesthesia, Epidural; Anesthesia, General

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General anesthesia (Active Comparator): Patients will receive general anesthesia
  Interventions: Procedure: general anesthesia
- Epidural anesthesia (Experimental): Patients will receive epidural anesthesia
  Interventions: Procedure: Epidural anesthesia

INTERVENTIONS:
Procedure: Epidural anesthesia — Segmental epidural analgesia
  Arms: Epidural anesthesia
Procedure: general anesthesia — general anesthesia
  Arms: General anesthesia

SUMMARY:
This study aim is to compare the efficiency and safety of segmental epidural block versus general anesthesia in cancer patients undergoing surgical feeding jejunostomy

DETAILED DESCRIPTION:
Comparing general anesthesia versus segmental epidural anesthesia in feeding jejunostomy

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for surgical feeding jejunostomy more than 18 years old

Exclusion Criteria:

* patien refusal Coagulation defect Abnormal kidney or liver functions Local infection at site of block Bone metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2021-04-25 (Actual); Study Completion 2021-04-26 (Actual)

PRIMARY OUTCOMES:
Analgesic requirements | first 24 hours
  Analgesic requirments
Haemodynamics | periooperative time
  blood pressure

SECONDARY OUTCOMES:
VAS score | 24 hours
  visual analouge scale 0 minimum to 10 maximum score

CONTACTS AND LOCATIONS:
Overall Officials: Walaa Y Elsabeeny, MD, Principal Investigator — Lecturer
Locations (1):
- National Cancer Institute, Cairo, Egypt